CLINICAL TRIAL: NCT02882152
Title: Continuous Femoral Nerve Blockade and Single Shot Sciatic Nerve Block Compared to Intrathecal Morphine for Total Knee Arthroplasty
Brief Title: Femoral/Sciatic Block for Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0257/09
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2014-09

CONDITIONS: Knee Injuries
Keywords: Analgesia; Nerve Block; Pain, Postoperative
MeSH Terms: conditions — Knee Injuries; Agnosia; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- femoral blockade (Experimental): femoral nerve blockade followed by a catheter placement for continuous infusion and a "single shot" block of the sciatic nerve
  Interventions: Procedure: femoral nerve blockade
- Morphine (Active Comparator): intrathecal morphine
  Interventions: Procedure: morphine

INTERVENTIONS:
Procedure: femoral nerve blockade — femoral nerve blockade followed by a catheter placement for continuous infusion and a "single shot" block of the sciatic nerve at the end of the surgery
  Arms: femoral blockade
Procedure: morphine — Intrathecal morphine injection
  Arms: Morphine

SUMMARY:
Knee arthroplasty has a high potential for postoperative pain. This study compares analgesia and postoperative bleeding from intrathecal morphine with the continuous femoral and a single-shot sciatic nerve blockades.

DETAILED DESCRIPTION:
This study aims to compare intrathecal morphine as a technique for analgesia with the femoral nerve blockade associated with a single-shot sciatic nerve blockade. Analgesic efficacy, the incidence of adverse effects, and postoperative bleeding were evaluated

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old, American Society of Anesthesiologists (ASA) physical status from I to III who underwent total knee arthroplasty

Exclusion Criteria:

* Patients aged below 18 years old, ASA IV or V physical status, infection near the puncture site, coagulation disorders, preexisting neurological disorders, allergy report to local anesthetics, pregnancy and lactation, contraindications to spinal block and refusal to sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Mansur, MD. PhD, Study Director — Comissão de Ética para Análise de Projetos de Pesquisa-CAPPesq - HCFMUSP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer MC, Pogatzki-Zahn EM, Zahn PK. Regional analgesia techniques for total knee replacement. Curr Opin Anaesthesiol. 2014 Oct;27(5):501-6. doi: 10.1097/ACO.0000000000000115. PMID 25111605
- [Background] Guay J, Kopp S. Epidural pain relief versus systemic opioid-based pain relief for abdominal aortic surgery. Cochrane Database Syst Rev. 2016 Jan 5;2016(1):CD005059. doi: 10.1002/14651858.CD005059.pub4. PMID 26731032
- [Background] Bujedo BM, Santos SG, Azpiazu AU. A review of epidural and intrathecal opioids used in the management of postoperative pain. J Opioid Manag. 2012 May-Jun;8(3):177-92. doi: 10.5055/jom.2012.0114. PMID 22798178
- [Background] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Background] Li XM, Huang CM, Zhong CF. Intrathecal morphine verse femoral nerve block for pain control in total knee arthroplasty: A meta-analysis from randomized control trials. Int J Surg. 2016 Aug;32:89-98. doi: 10.1016/j.ijsu.2016.06.043. Epub 2016 Jul 6. PMID 27370542
- [Background] Kadic L, Boonstra MC, DE Waal Malefijt MC, Lako SJ, VAN Egmond J, Driessen JJ. Continuous femoral nerve block after total knee arthroplasty? Acta Anaesthesiol Scand. 2009 Aug;53(7):914-20. doi: 10.1111/j.1399-6576.2009.01965.x. Epub 2009 Apr 15. PMID 19388886
- [Background] Grape S, Kirkham KR, Baeriswyl M, Albrecht E. The analgesic efficacy of sciatic nerve block in addition to femoral nerve block in patients undergoing total knee arthroplasty: a systematic review and meta-analysis. Anaesthesia. 2016 Oct;71(10):1198-209. doi: 10.1111/anae.13568. Epub 2016 Jul 29. PMID 27469381
- [Background] Raj PP, Parks RI, Watson TD, Jenkins MT. A new single-position supine approach to sciatic-femoral nerve block. Anesth Analg. 1975 Jul-Aug;54(4):489-93. doi: 10.1213/00000539-197507000-00020. PMID 1170786
- [Derived] Alvarez NER, Ledesma RJG, Hamaji A, Hamaji MWM, Vieira JE. Continuous femoral nerve blockade and single-shot sciatic nerve block promotes better analgesia and lower bleeding for total knee arthroplasty compared to intrathecal morphine: a randomized trial. BMC Anesthesiol. 2017 May 12;17(1):64. doi: 10.1186/s12871-017-0355-x. PMID 28499420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Femoral Blockade | Morphine
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Blockade | Morphine | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.3) | 58.3 (10.5) | 62.5 (10.3)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 3 | 6 | 9
Weight [Mean (Standard Deviation); unit: kg] | 70.7 (20.0) | 77.5 (16.9) | 76.6 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Efficacy
Description: Pain with verbal numeric rating scale (VNRS). VNRS has 11 points, from zero to 10 (zero= no pain, 1-3 = mild pain, 4-5 = moderate pain, 7-9 = severe pain, 10 = unbearable pain).
Time Frame: baseline (zero hour: discharge of post-anesthesia care unit-PACU), 24hs, 48hs, 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Blockade | Morphine
Number analyzed (Participants) | 19 | 20
units on a scale
  Zero hour (discharge of PACU) | 0 (0) | 0.1 (0.1)
  24 hours | 0.6 (0.2) | 3.0 (0.5)
  48 hours | 0.3 (0.1) | 3.5 (0.4)
  72 hours | 0.1 (0.1) | 2.6 (0.3)
Statistical Analysis 1: Comparison: Femoral Blockade vs Morphine; Results were compared by means of the ANOVA of repeated measures followed by Bonferroni test. Comparing: all four moments, from zero to 72hs within femoral blockade group, all four moments within morphine group, and all four moments between the groups; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Postoperative Bleeding
Description: Postoperative bleeding volume (ml)
Time Frame: baseline (discharge of post-anesthesia care unit-PACU), 24hs, 48hs, 72 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Femoral Blockade | Morphine
Number analyzed (Participants) | 19 | 20
mL
  Zero hour (discharge of PACU) | 136.5 (20.5) | 271.8 (33.3)
  24 hours | 180.5 (19.7) | 334.7 (39.6)
  48 hours | 69.2 (20.7) | 111.9 (28.4)
  72 hours | 20.0 (0.0) | 155.3 (39.1)
Statistical Analysis 1: Comparison: Femoral Blockade vs Morphine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: baseline (zero hour: discharge of post-anesthesia care unit-PACU), 24hs, 48hs, 72 hours
Description: pruritus, nausea and vomiting. All patients were observed by an anesthesiologists during post-anesthesia care unit (PACU) for these events, and interviewed by an anesthesiologist for report or register of these events at 24hs, 48hs, and 72 hours after PACU discharge
Arm/Group | Femoral Blockade | Morphine
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes